CLINICAL TRIAL: NCT00854100
Title: A Double-Blind, Placebo-Controlled Study of Cariprazine (RGH-188) As Adjunctive Therapy In Major Depressive Disorder
Brief Title: Safety and Efficacy of Cariprazine As Adjunctive Therapy In Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGH-MD-71; NCT03605784 (obsolete NCT alias)
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Major Depressive Disorder
Keywords: Adjunctive; Depression; Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Antidepressive Agents; cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Drug: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR) + Placebo
  Interventions: Drug: Antidepressant + placebo
- Cariprazine 0.1 - 0.3 mg (Experimental): Drug: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR)+ cariprazine low dose
  Interventions: Drug: Antidepressant + cariprazine (0.1-0.3 mg/day)
- Cariprazine 1.0 - 2.0 mg (Experimental): Drug: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR) + cariprazine high dose
  Interventions: Drug: Antidepressant + cariprazine (1-2 mg/d)

INTERVENTIONS:
Drug: Antidepressant + placebo — Drug: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR) + Placebo Oral, once daily for 8 weeks following an 8 week Prospective Treatment (Baseline) Period.
  Arms: Placebo
Drug: Antidepressant + cariprazine (0.1-0.3 mg/day) — Drug: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR) + cariprazine (0.1-0.3 mg/d) Oral, once daily for 8 weeks following an 8 week Prospective Treatment (Baseline) Period.
  Arms: Cariprazine 0.1 - 0.3 mg
Drug: Antidepressant + cariprazine (1-2 mg/d) — Drug: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR) + cariprazine (1-2 mg/d) Oral, once daily for 8 weeks following an 8 week Prospective Treatment (Baseline) Period.
  Arms: Cariprazine 1.0 - 2.0 mg

SUMMARY:
This is an outpatient study to evaluate the safety, and efficacy of RGH-188 as an add-on therapy to standard antidepressants in patients who did not respond to previous antidepressant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-65 years old
* Currently meet the DSM-IV-TR criteria for moderate to severe MDD without psychotic features.
* Previous failure to respond to adequate trials of one or two ADTs with less than 50% reduction in depressive symptoms during the present episode.

Exclusion Criteria:

* DSM-IV-TR based diagnosis of an axis I disorder, other than MDD, or any axis I disorder other than MDD that was the primary focus of treatment within 6 months before Visit 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2009-06-30 (Actual); Primary Completion 2010-12-06 (Actual); Study Completion 2010-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hayes, PhD, Study Director — Forest Laboratories
Locations (40):
- United States (40):
  - Forest Investigative Site 040, Phoenix, Arizona
  - Forest Investigative Site 038, Scottsdale, Arizona
  - Forest Investigative Site, Arcadia, California
  - Forest Investigative Site, Encino, California
  - Forest Investigative Site, Garden Grove, California
  - Forest Investigative Site, Irvine, California
  - Forest Investigative Site 013, Los Alamitos, California
  - Forest Investigative Site 041, National City, California
  - Forest Investigative Site, Oceanside, California
  - Forest Investigative Site 025, Denver, Colorado
  - Forest Investigative Site, Norwich, Connecticut
  - Forest Investigative Site, Washington D.C., District of Columbia
  - Forest Investigative Site 007, Jacksonville, Florida
  - Forest Investigative Site 012, West Palm Beach, Florida
  - Forest Investigative Site 033, Atlanta, Georgia
  - Forest Investigative Site, Roswell, Georgia
  - Forest Investigative Site, Overland Park, Kansas
  - Forest Investigative Site 042, Fall River, Massachusetts
  - Forest Investigative Site 034, Pittsfield, Massachusetts
  - Forest Investigative Site, Omaha, Nebraska
  - Forest Investigative Site, Cherry Hill, New Jersey
  - Forest Investigative Site 043, Brooklyn, New York
  - Forest Investigative Site 020, Mount Kisco, New York
  - Forest Investigative Site 039, New York, New York
  - Forest Investigative Site 029, New York, New York
  - Forest Investigative Site 001, The Bronx, New York
  - Forest Investigative Site 032, Raleigh, North Carolina
  - Forest Investigative Site, Canton, Ohio
  - Forest Investigative Site, Dayton, Ohio
  - Forest Investigative Site 015, Portland, Oregon
  - Forest Investigative Site 006, Media, Pennsylvania
  - Forest Investigative Site, Philadelphia, Pennsylvania
  - Forest Investigative Site 023, Memphis, Tennessee
  - Forest Investigative Site 031, Memphis, Tennessee
  - Forest Investigative Site, Nashville, Tennessee
  - Forest Investigative Site, San Antonio, Texas
  - Forest Investigative Site, Woodstock, Vermont
  - Forest Investigative Site, Richmond, Virginia
  - Forest Investigative Site, Bellevue, Washington
  - Forest Investigative Site, Seattle, Washington

REFERENCES:
- [Derived] Fava M, Durgam S, Earley W, Lu K, Hayes R, Laszlovszky I, Nemeth G. Efficacy of adjunctive low-dose cariprazine in major depressive disorder: a randomized, double-blind, placebo-controlled trial. Int Clin Psychopharmacol. 2018 Nov;33(6):312-321. doi: 10.1097/YIC.0000000000000235. PMID 30045066

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The randomized population for RGH-MD-71 totaled 231 participants
Groups:
- Cariprazine 0.1 - 0.3 mg: Drug: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR) + cariprazine low dose
Period: Overall Study
Arm/Group | Placebo | Cariprazine 0.1 - 0.3 mg | Cariprazine 1.0 - 2.0 mg
Started | 81 | 76 | 74
Completed | 72 | 70 | 63
Not Completed | 9 | 6 | 11
Not completed — Inability to complete the study visits | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Protocol Violation | 2 | 4 | 3
Not completed — Adverse Event | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: A total of 231 patients were eligible for randomization to double-blind treatment; 230 patients were randomized and received at least 1 dose of treatment (Double-blind Safety Population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine 0.1 - 0.3 mg | Cariprazine 1.0 - 2.0 mg | Total
Number analyzed (Participants) | 81 | 76 | 73 | 230
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.2 (10.2) | 46.6 (11.7) | 44.2 (12.1) | 45.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 52 | 51 | 164
  Male | 20 | 24 | 22 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 9 | 25
  Not Hispanic or Latino | 74 | 67 | 64 | 205
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 15 | 11 | 36
  White | 69 | 57 | 60 | 186
  More than one race | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The patient is rated on a scale from 0-6 on 10 items. Apparent sadness, reported sadness, lassitude, pessimistic thoughts, inner tension, suicidal thoughts, reduced sleep and appetite, concentration difficulties, inability to feel. The overall MADRS score ranges from 0-60, with 0 meaning no symptoms and score of 60 meaning maximum severity. The primary efficacy parameter was the change in MADRS score totals from the scores taken at Baseline (Week 8) and during at least one more time point up to and including Week 16.
Time Frame: Baseline (Week 8) to Week 16
Population: 231 patients were randomized, and of them, 230 received at least 1 dose of treatment (Double-blind Safety Population), and had at least a baseline and 1 post-baseline MADRS assessment (Double-blind Intent To Treat Population). All patients in the Double-blind Intent To Treat Population were included in the efficacy analyses.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Cariprazine 0.1 - 0.3 mg | Cariprazine 1.0 - 2.0 mg
Number analyzed (Participants) | 81 | 76 | 73
Units on a Scale | -8.0 (1.0) | -7.5 (1.1) | -9.8 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 0.1 - 0.3 mg; Test type: Superiority; p = 0.746, ANCOVA; Least Squares Mean Difference = 0.5, 95% CI 2-sided [-2.4 to 3.4]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 1.0 - 2.0 mg; Test type: Superiority; p = 0.227, ANCOVA; Least Squares Mean Difference = -1.8, 95% CI 2-sided [-4.8 to 1.1]

2. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I)
Description: The Clinical Global Impression-Improvement (CGI-I) scale is a clinician rated scale that, in this study, will be used to rate total improvement or worsening of mental illness starting at Visit 2 (Week 2) and taken at every visit through Visit 11 (Week 16). The patient will be rated on a scale from 1 to 7, 1 indicating that the patient is very much improved and 7 indicating that the patient is very much worse. The secondary efficacy parameter was the CGI-I total score at Week 16.
Time Frame: Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Cariprazine 0.1 - 0.3 mg | Cariprazine 1.0 - 2.0 mg
Number analyzed (Participants) | 81 | 76 | 73
Units on a Scale | 2.5 (0.1) | 2.5 (0.1) | 2.3 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 0.1 - 0.3 mg; Test type: Superiority; p = 0.918, ANCOVA; Least Squares Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 1.0 - 2.0 mg; Test type: Superiority; p = 0.167, ANCOVA; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.1]

ADVERSE EVENTS:
Time Frame: Up to 20 weeks
Description: Any AE includes the prospective ADT lead-in, double-blind treatment and 30 -day safety follow up will be considered a treatment-emergent adverse event (TEAE). A TEAE that occurs more than 30 days after the last dose of the investigational product will not be summarized for the safety follow-up period.1 patient left the study after they were randomized to the Cariprazine 1.0-2.0 mg arm, but never took the drug. Therefore, that patient is only captured in the lead in period data.
Groups:
- Prospective Antidepressant-Therapy Lead In Period: Interventions included: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR) for 8 weeks prior to randomization
- Placebo: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR) + Placebo for 8 weeks. AE reporting covers this 8 week period plus the 30 day safety follow up that proceeds it.
- Cariprazine 0.1 - 0.3 mg: Drug: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR) + cariprazine low dose for 8 weeks. AE reporting covers this 8 week period plus the 30 day safety follow up that proceeds it.
- Cariprazine 1.0 - 2.0 mg: Drug: Antidepressant (citalopram, duloxetine, escitalopram, sertraline, or venlafaxine XR) + cariprazine high dose for 8 weeks. AE reporting covers this 8 week period plus the 30 day safety follow up that proceeds it.
Arm/Group | Prospective Antidepressant-Therapy Lead In Period | Placebo | Cariprazine 0.1 - 0.3 mg | Cariprazine 1.0 - 2.0 mg
All-Cause Mortality (participants affected / at risk) | 1/502 | 0/81 | 0/76 | 0/73
Serious Adverse Events (participants affected / at risk) | 9/502 | 1/81 | 0/76 | 1/73
Other Adverse Events (participants affected / at risk) | 262/502 | 32/81 | 29/76 | 35/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Antidepressant-Therapy Lead In Period (N=502) | Placebo (N=81) | Cariprazine 0.1 - 0.3 mg (N=76) | Cariprazine 1.0 - 2.0 mg (N=73)
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Serotonin Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alcohol Abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Homicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Chronic Obstructive Pulmanary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective Antidepressant-Therapy Lead In Period (N=502) | Placebo (N=81) | Cariprazine 0.1 - 0.3 mg (N=76) | Cariprazine 1.0 - 2.0 mg (N=73)
Headache (Nervous system disorders) | 73 | 3 | 8 | 6
Dizziness (Nervous system disorders) | 31 | 7 | 4 | 6
Fatigue (General disorders) | 36 | 3 | 2 | 5
Insomnia (Psychiatric disorders) | 60 | 3 | 2 | 7
Nasopharyngitis (Infections and infestations) | 0 | 5 | 1 | 6
Nausea (Gastrointestinal disorders) | 70 | 5 | 5 | 5
Dry Mouth (Gastrointestinal disorders) | 53 | 1 | 2 | 4
Constipation (Gastrointestinal disorders) | 35 | 1 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 36 | 5 | 4 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 29 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 25 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 3 | 2 | 4
Tremor (Nervous system disorders) | 0 | 4 | 0 | 4
Anxiety (Psychiatric disorders) | 0 | 3 | 1 | 4
Restlessness (Psychiatric disorders) | 0 | 1 | 1 | 7
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc